CLINICAL TRIAL: NCT00299962
Title: A Phase I Clinical Trial of Repeated Dose Intrapleural Adenoviral-Mediated Interferon-beta (BG00001, Ad.hIFN-β for Pleural Malignancies
Brief Title: Gene Therapy for Pleural Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803776; P01CA066726 (NIH)
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Pleural Mesothelioma; Metastatic Pleural Effusions
Keywords: gene therapy; immunotherapy
MeSH Terms: conditions — Mesothelioma, Malignant; Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose level 4 (Experimental)
  Interventions: Biological: Adenoviral-mediated Interferon-beta; Biological: SCH 721015
- Dose level 5 (Experimental)
  Interventions: Biological: Adenoviral-mediated Interferon-beta; Biological: SCH 721015
- Dose Level 1 (Experimental): on Days 1 and 15
  Interventions: Biological: SCH 721015
- Dose Level 2 (Experimental): On Days 1 and 15
  Interventions: Biological: SCH 721015
- Dose Level 3 (Experimental): On Days 1 and 15
  Interventions: Biological: SCH 721015

INTERVENTIONS:
Biological: Adenoviral-mediated Interferon-beta — BG00001 at doses 1.5 x 10e12 and 3 x 10e12 viral particles Days 1 and 8
  Arms: Dose level 4; Dose level 5
Biological: SCH 721015 — Comparison of different doses and frequency of investigational agent
  Other Names: Adenoviral-mediated Interferon-beta; Ad.hIFN-beta

SUMMARY:
This Phase I study will evaluate the safety of two doses of BG00001 at different doses and intervals. Eligible subjects will have:

* malignant pleural mesothelioma, or
* pleural effusions who have progressed through at least one prior therapy or have refused therapy

BG00001 is given twice through a catheter in the pleural space.

DETAILED DESCRIPTION:
Ad.hIFN-β (BG00001) is a replication-defective recombinant adenoviral vector containing the human interferon-beta (hIFN-β) gene. This Phase I study is designed to evaluate the safety and maximum tolerated dose (MTD) of two doses of intrapleural (IP) Ad.hIFN-β in subjects with pleural malignancies either metastatic or pleural mesothelioma.

Five dose levels will be studied:

* Dose levels 1, 2, and 3 will be given on Days 1 and 15
* Dose levels 4 and 5 will be given on Days 1 and 8

ELIGIBILITY:
Inclusion Criteria:

* must have malignant pleural effusion from mesothelioma or metastatic from primary lung, breast, gastrointestinal, genitourinary, melanoma, or sarcoma
* must have evaluable disease
* must have ECOG performance status of 2
* must have pleural space involved with tumor accessible for pleural catheter
* must have FEV1 > 1 liter or 40% of predicted value
* must have completed radiotherapy and/or treatment with chemotherapy, cytotoxic, or immunologic agents 4 weeks prior to dosing with BG00001
* concurrent Tarceva is allowed if patients has been on a stable dose for at least three months and has not had serious adverse events
* patients on stable dose of hormone may continue use of hormone
* patients on stable dose of Tarceva for 3 months and without complications may remain on Tarceva

Exclusion Criteria:

* malignant pleural effusions secondary to lymphoma
* rapidly re-accumulating, symptomatic malignant pleural effusions that require immediate mechanical or chemical pleurodesis for palliation
* untreated brain metastases
* use of concurrent systemic steroids or immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-03; Primary Completion 2008-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine toxicity of two doses of intrapleural BG00001 (Ad.hIFN-β over 8 days, and | Through Day 85

SECONDARY OUTCOMES:
To assess systemic and intrapleural cytokine responses as well as cellular and humoral immune responses after repeated BG00001 instillation, | Through Day 85
and to assess, in a preliminary way, efficacy via tumor regression, time to progression and survival. | 15 years or until subject dies, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Sterman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: mesothelioma research foundation — http://www.marf.org